CLINICAL TRIAL: NCT02337907
Title: A Multi-centre, Double-blind, Parallel-group, Randomised Controlled Study to Investigate Efficacy, Safety and Tolerability of Orally Administered BI 409306 During a 12-week Treatment Period Compared to Placebo in Patients With Cognitive Impairment Due to Alzheimer's Disease
Brief Title: BI 409306 in Patients With Cognitive Impairment Due to Alzheimer's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.7; 2013-005040-28 (EudraCT Number)
Record Dates: First submitted 2014-12-23; First posted 2015-01-14 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BI 409306; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 409306 dose 1 (Experimental)
  Interventions: Drug: Placebo; Drug: BI 409306
- BI 409306 dose 2 (Experimental)
  Interventions: Drug: Placebo; Drug: BI 409306
- BI 409306 dose 3 (Experimental)
  Interventions: Drug: Placebo; Drug: BI 409306
- Active Comparator Donepezil (Active Comparator)
  Interventions: Drug: Placebo; Drug: Donepezil
- BI 409306 dose 4 (Experimental)
  Interventions: Drug: Placebo; Drug: BI 409306

INTERVENTIONS:
Drug: Placebo — for blinding purposes
Drug: Placebo
  Arms: Placebo comparator
Drug: BI 409306
  Arms: BI 409306 dose 1; BI 409306 dose 2; BI 409306 dose 3; BI 409306 dose 4
Drug: Donepezil
  Arms: Active Comparator Donepezil

SUMMARY:
The study is designed to compare the effects of BI 409306 compared to placebo in patients with cognitive impairment due to Alzheimer's Disease

ELIGIBILITY:
Inclusion criteria:

* Patients with early signs of dementia of Alzheimer Type
* Male and female patients with an age of at least 55 years
* Previous use of Alzheimer's Disease (AD) medications (AChEIs, memantine) is allowed up 3 month prior to screening. Patients who are currently taking AChEIs are eligible as long as they have been using a stable dose for at least 3 months prior to screening and no change is foreseen for the duration of the study. This dose must be consistent with the product label in the concerned country. Patients currently taking memantine are excluded.
* Patients must have at least 6 years of formal education and fluency in the test language as verbally confirmed by the patient and documented by the study investigator.
* Patients must have a reliable study partner (per investigator judgement, for instance a family member, partner etc., guardian or, if applicable, a legal representative)

Exclusion criteria:

* Cognitive impairment or dementia with any etiology other than Alzheimer's Disease (AD)
* Substantial concomitant cerebrovascular disease (defined by a history of a stroke / intracranial haemorrhagia) temporally related to the onset of worsening of cognitive impairment per investigator judgement
* Medical history or diagnosis of any of symptomatic and unstable/uncontrolled conditions per investigator judgement
* Any other psychiatric disorders such as schizophrenia, or mental retardation
* Previous participation in investigational drug studies of mild cognitive impairment/Dementia of Alzheimer Type (DAT) within three months prior to screening. Having received active treatment in any other study targeting disease modification of AD like Aß immunization and tau therapies. Previous participation in studies with non-prescription medications, vitamins or other nutritional formulations is allowed.
* Clinically significant uncompensated hearing loss in the judgment of the investigator. Use of hearing aids is allowed.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (60):
- United States (10):
  - California Neuroscience Research, Sherman Oaks, California
  - Bioclinica Research, Orlando, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Indiana University, Indianapolis, Indiana
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Psychiatry And Alzheimer's Care of Rochester, PLLC, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - ANI Neurology, PLLC, dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - The Memory Clinic, Bennington, Vermont
- Private Practice for Psychiatry and Neurology, Vienna, Austria
- Belgium (4):
  - Brussels-UNIV Brugmann -Horta, Brussels
  - AZ Sint-Blasius, Dendermonde
  - UNIV UZ Gent, Ghent
  - Mons - UNIV Ambroise Paré, Mons
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - Pasqua Hospital, Regina, Saskatchewan
  - Institut universitaire de geriatrie Sherbrooke, Québec
- France (7):
  - HOP Pellegrin, Bordeaux
  - HOP Bocage, Dijon
  - HOP Timone, Marseille
  - HOP Gui de Chauliac, Montpellier
  - HOP Nord Laënnec, Nantes
  - HOP La Pitié Salpêtrière, Paris
  - HOP Jean Bernard, Géria, Poitiers, Poitiers
- Germany (9):
  - Praxis Dr. med. Volker Schumann, Berlin
  - emovis GmbH, Berlin
  - St. Josef- und St. Elisabeth-Hospital gGmbH, Bochum
  - Neuro Centrum Science GmbH, Erbach im Odenwald
  - AFL Arzneimittelforschung Leipzig GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Universitätsklinikum Ulm, Ulm
  - Neurologie und Psychiatrie / Psychotherapie, Westerstede
- Italy (3):
  - P.O. Bellaria IRCCS Istituto delle scienze Neurologiche di Bologna, Bologna
  - Azienda Ospedaliera Careggi, Florence
  - Azienda Ospedaliera di Parma, Parma
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
- Poland (8):
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Mental Health Center Biomed, Kielce
  - Non-Public Outpatient Clinic Neuromed M. i M. Nastaj, Lublin
  - Inst. of Rural Health, Spec. Outp. Clin. & Rural Occup. Dis., Lublin
  - Non-Public Outpatient Clinic Neuro-Kard Ilkowski & Partners, Poznan
  - Medical Center Senior, Sopot
  - EUROMEDIS Sp. z o.o., Szczecin, Szczecin
  - Reg. Specialist Hospital Wroclaw, Research & Develop. Center, Wroclaw
- Portugal (8):
  - Hospital Fernando Fonseca, EPE, Amadora
  - Hospital de Braga-Escala Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Hospital Senhora Oliveira Guimarães,EPE, Guimarães
  - CHLO, EPE - Hospital Egas Moniz, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - ULSM, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
- United Kingdom (4):
  - Royal United Hospital, Bath
  - Ninewells Hospital & Medical School, Dundee, Scotland
  - West Devon (Tavistock) CMHT & Memory Clinic (EDI), Ivybridge
  - Re-Cognition Health, Plymouth

REFERENCES:
- [Derived] Frolich L, Wunderlich G, Thamer C, Roehrle M, Garcia M Jr, Dubois B. Evaluation of the efficacy, safety and tolerability of orally administered BI 409306, a novel phosphodiesterase type 9 inhibitor, in two randomised controlled phase II studies in patients with prodromal and mild Alzheimer's disease. Alzheimers Res Ther. 2019 Feb 12;11(1):18. doi: 10.1186/s13195-019-0467-2. PMID 30755255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase II, multi-centre, double-blind, parallel-group, randomised, placebo controlled trial with patients with mild Alzheimer's disease. The randomisation allocation ratio was 1:1:1:1:2 of 10 milligram (mg), 25 mg, 50 mg once daily (QD), 25 mg twice a day (BID) of BI 409306 and placebo respectively.
Pre-assignment Details: All patients were screened for eligibility. All patients eligible after screening underwent a 2-week single-blind placebo run-in period before randomisation. Patients were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- BI 409306 10 Milligram (mg) Once Daily (QD): Patients were administered orally a tablet of 10 mg BI 409306 once daily for 12 weeks.
- BI 409306 25 mg QD: Patients were administered orally a tablet of 25 mg BI 409306 once daily for 12 weeks.
- BI 409306 50 mg QD: Patients were administered orally a tablet of 50 mg BI 409306 once daily for 12 weeks.
- BI 409306 25 mg Twice Daily (BID): Patients were administered orally a tablet of 25 mg BI 409306 twice daily for 12 weeks.
- Placebo Matching BI 409306: Patients were administered orally tablet of Placebo matching BI 409306 once daily for 12 weeks.
- Donepezil QD: Patients were administered orally over capsulated tablet of Donepezil once daily for 12 weeks.
Period: Overall Study
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306 | Donepezil QD
Started | 55 | 53 | 55 | 55 | 106 | 5
Completed | 51 | 49 | 54 | 51 | 96 | 4
Not Completed | 4 | 4 | 1 | 4 | 10 | 1
Not completed — Other than listed | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 2 | 5 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) included all patients who were randomised and treated with at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306 | Donepezil QD | Total
Number analyzed (Participants) | 55 | 53 | 55 | 55 | 106 | 5 | 329
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented.
  Years | 73.7 (8.4) | 74.2 (7.8) | 73.0 (6.5) | 74.8 (9.1) | 74.0 (7.7) | 79.6 (7.0) | 74.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female.
  Participants
    Female | 26 | 30 | 26 | 30 | 48 | 3 | 163
    Male | 29 | 23 | 29 | 25 | 58 | 2 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for ethnicity data.
  Participants
    Hispanic or Latino | 2 | 2 | 4 | 2 | 2 | 1 | 13
    Not Hispanic or Latino | 53 | 51 | 51 | 53 | 104 | 4 | 316
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 1 | 0 | 0 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 3 | 0 | 3
    White | 54 | 53 | 54 | 55 | 103 | 5 | 324
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neuropsychological Test Battery in Total Z-score After 12-week Treatment.
Description: Neuropsychological Test Battery (NTB) response, defined as change from baseline in total z-score after 12 weeks of treatment. The NTB consists of 9 validated components. Raw scores on each of the 9 NTB tests were converted to z-scores using the baseline means and standard deviations (SDs) for each test. The resultant z-scores were averaged to obtain a total z-score, incorporating all 9 NTB tests. The NTB Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean at baseline. Negative numbers indicate values lower than baseline and positive numbers indicate values higher than baseline. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: The full analysis set (FAS): FAS includes all randomised patients who were treated with at least one dose of trial medication and had a baseline and at least one post-baseline on-treatment primary endpoint NTB or secondary endpoint assessment. Observed cases (OC)
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- Pooled BI 409306: Patients were administered orally a tablet of BI 409306 (10 mg, 25 mg, 50 mg once daily and 25 mg twice daily)for 12 weeks.
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Pooled BI 409306 | Placebo Matching BI 409306
Number analyzed (Participants) | 54 | 50 | 55 | 55 | 214 | 101
Z-score | 0.13 (0.059) | 0.17 (0.061) | 0.16 (0.056) | 0.01 (0.060) | 0.12 (0.30) | 0.15 (0.045)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; Mixed Model Repeated Measurement (MMRM) includes fixed, categorical effects of treatment, visit, current Acetylcholine Esterase Inhibitor (AChEI) use (Yes, No), and treatment-by-visit interaction, as well as the continuous fixed covariates of baseline, and baseline-by-visit interaction; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.7907, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.163 to 0.124], Standard Error of Mean 0.073 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.7622, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.125 to 0.171], Standard Error of Mean 0.075 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.8789, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.130 to 0.152], Standard Error of Mean 0.071 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.0609, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.285 to 0.006], Standard Error of Mean 0.074 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 5: Comparison: Pooled BI 409306 vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — H1-0: Mean NTB response of pooled doses of 10 mg QD, 25 mg QD, 25 mg BID and 50 mg QD = Mean NTB response of placebo; p = 0.5687, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.135 to 0.074], Standard Error of Mean 0.053 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

2. Primary Outcome: Change From Baseline in Neuropsychological Test Battery in Total Z-score After 12-week Treatment From Two Sister Trials, Present 1289.5 (NCT02240693) and 1289.7 (NCT02337907)
Description: Neuropsychological Test Battery (NTB) response, defined as change from baseline in total z-score after 12 weeks of treatment. The NTB consists of 9 validated components. Raw scores on each of the 9 NTB tests were converted to z-scores using the baseline means and standard deviations (SDs) for each test. The resultant z-scores were averaged to obtain a total z-score, incorporating all 9 NTB tests. The NTB Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean at baseline. Negative numbers indicate values lower than baseline and positive numbers indicate values higher than baseline. The number of low test scores decreased with higher levels of intellectual abilities. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS (OC) and for pooled group FAS
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Pooled BI 409306 | Placebo Matching BI 409306
Number analyzed (Participants) | 76 | 71 | 76 | 76 | 299 | 144
Z-score | 0.20 (0.046) | 0.19 (0.048) | 0.19 (0.046) | 0.10 (0.047) | 0.17 (0.025) | 0.19 (0.035)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; Mixed Model Repeated Measurement (MMRM) includes fixed, categorical effects of treatment, visit, current Acetylcholine Esterase Inhibitor (AChEI) use (Yes, No), and treatment-by-visit interaction, as well as the continuous fixed covariates of baseline, and baseline-by-visit interaction. The study identifier is also a categorical covariate for the twin studies analyses; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.8694, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.101 to 0.120], Standard Error of Mean 0.056 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.9512, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.116 to 0.109], Standard Error of Mean 0.057 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.9321, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.105 to 0.115], Standard Error of Mean 0.056 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — H0: The dose group with the peak response in the respective model Mean NTB response = Mean NTB response of placebo; p = 0.1288, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.199 to 0.025], Standard Error of Mean 0.057 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 5: Comparison: Pooled BI 409306 vs Placebo Matching BI 409306; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — H1-0: Mean NTB response of pooled doses of 10 mg QD, 25 mg QD, 25 mg BID and 50 mg QD = Mean NTB response of placebo; p = 0.6492, Mixed Model Repeated Measurement (MMRM) — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.098 to 0.061], Standard Error of Mean 0.041 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS-ADL) Total Score After 12-week Treatment
Description: Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS-ADL) is a rating scale used to assess basic and instrumental activities of daily living. In the full version of the scale, 23 items are rated by the investigator using information supplied by the caregiver. Each item has a score range varying from 0-3 to 0-5. The sum score can range from 0 to 78. Higher scores indicate better function. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Number analyzed (Participants) | 54 | 50 | 55 | 55 | 101
Unit on scale | 0.10 (0.853) | -0.99 (0.892) | 0.35 (0.847) | -1.07 (0.855) | -0.58 (0.639)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; The dependent variable was the change from the baseline score at Week 12. The model included fixed, categorical covariates of treatment as well as fixed continuous covariates of baseline score; Test type: Superiority — Analyses of covariance (ANCOVA) were used to assess between-group differences in the modelled changes from baseline to Week 12; p = 0.5287, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-1.43 to 2.77], Standard Error of Mean 1.066 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.7105, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-2.57 to 1.76], Standard Error of Mean 1.099 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.3822, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-1.16 to 3.03], Standard Error of Mean 1.064 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.6472, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-2.59 to 1.61], Standard Error of Mean 1.066 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

4. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) Total Score After 12-week Treatment
Description: The CDR-SB is obtained through semi-structured interviews of patients and informants, and cognitive functioning was rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Each domain was rated on a 5-point scale of functioning as follows: 0-no impairment; 0.5-questionable impairment; 1-mild impairment; 2-moderate impairment and 3-severe impairment. Only personal care was scored on a 4-point scale without a 0.5 rating available. The higher the score, the greater the severity of dementia. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Number analyzed (Participants) | 54 | 50 | 55 | 55 | 101
Unit on scale | 0.1 (0.23) | 0.3 (0.23) | 0.1 (0.21) | 0.2 (0.22) | 0.1 (0.16)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7551, Mixed-effects Model for Repeated Measure — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.46 to 0.64], Standard Error of Mean 0.28 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3643, Mixed-effects Model for Repeated Measure — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.29 to 0.80], Standard Error of Mean 0.28 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7822, Mixed-effects Model for Repeated Measure — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.45 to 0.60], Standard Error of Mean 0.27 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6889, Mixed-effects Model for Repeated Measure — p-value was nominal and not adjusted; Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.43 to 0.65], Standard Error of Mean 0.28 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

5. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog11) Total Score After 12-week Treatment
Description: Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog11) is an 11-item cognitive subscale that objectively measures memory, language, orientation, and praxis with a total score range of 0 to 70. The greater the dysfunction, the greater the score. Least Squares Mean is actually an adjusted mean change from baseline.
Time Frame: Baseline and 12 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306
Number analyzed (Participants) | 54 | 50 | 55 | 55 | 101
Unit on scale | 1.14 (0.738) | 0.94 (0.776) | 1.11 (0.746) | 2.29 (0.746) | -0.18 (0.568)
Statistical Analysis 1: Comparison: BI 409306 10 Milligram (mg) Once Daily (QD) vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1595, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [-0.52 to 3.15], Standard Error of Mean 0.933 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 2: Comparison: BI 409306 25 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.2455, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-0.77 to 3.01], Standard Error of Mean 0.962 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 3: Comparison: BI 409306 50 mg QD vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1732, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [-0.57 to 3.13], Standard Error of Mean 0.940 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences
Statistical Analysis 4: Comparison: BI 409306 25 mg Twice Daily (BID) vs Placebo Matching BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0088, ANCOVA — p-value was nominal and not adjusted; Mean Difference (Final Values) = 2.47, 95% CI 2-sided [0.63 to 4.31], Standard Error of Mean 0.936 — The mean difference is actually adjusted mean of difference and the dispersion value is standard error of differences

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 7 days after last administration of BI 409306, up to 16 weeks.
Description: The treated set (TS) used (all patients who were randomised and treated with at least one dose of trial medication.) for safety assessment.
Arm/Group | BI 409306 10 Milligram (mg) Once Daily (QD) | BI 409306 25 mg QD | BI 409306 50 mg QD | BI 409306 25 mg Twice Daily (BID) | Placebo Matching BI 409306 | Donepezil QD
All-Cause Mortality (participants affected / at risk) | 1/55 | 0/53 | 0/55 | 0/55 | 0/106 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/55 | 3/53 | 1/55 | 3/55 | 8/106 | 0/5
Other Adverse Events (participants affected / at risk) | 6/55 | 9/53 | 7/55 | 2/55 | 8/106 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 10 Milligram (mg) Once Daily (QD) (N=55) | BI 409306 25 mg QD (N=53) | BI 409306 50 mg QD (N=55) | BI 409306 25 mg Twice Daily (BID) (N=55) | Placebo Matching BI 409306 (N=106) | Donepezil QD (N=5)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 10 Milligram (mg) Once Daily (QD) (N=55) | BI 409306 25 mg QD (N=53) | BI 409306 50 mg QD (N=55) | BI 409306 25 mg Twice Daily (BID) (N=55) | Placebo Matching BI 409306 (N=106) | Donepezil QD (N=5)
Nasopharyngitis (Infections and infestations) | 1 | 4 | 3 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 2 | 5 | 1 | 1 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
There were 5 patients who were randomised to donepezil arm which was dropped from the trial with protocol amendment. No further patients were randomised to this arm, but patients already randomised continued in the trial as originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02337907/SAP_000.pdf
  • Study Protocol (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT02337907/Prot_001.pdf